CLINICAL TRIAL: NCT03357926
Title: SAFE-ME - Prospective Database for Prediction of Atrial Fibrillation in Pacemaker and ICD Patients
Brief Title: Prospective Database for Prediction of Atrial Fibrillation in Pacemaker and ICD Patients
Acronym: SAFE-ME
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 29-229 ex 16/17
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Pacemaker Ddd; ICD
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation Group
  Interventions: Diagnostic Test: 24 hour Holter ECG Monitoring

INTERVENTIONS:
Diagnostic Test: 24 hour Holter ECG Monitoring — 24 hour Holter ECG Monitoring

SUMMARY:
Atrial fibrillation (AF) is associated with a five-fold increased risk of cerebrovascular stroke. While the risk of stroke in patients with known AF can be calculated via AF stroke prediction risk scores, the prediction of AF occurrence per se in individual patients remains difficult.

We will recruit 250 patients with an implanted dual-chamber Pacemaker (PM) or an implantable cardioverter Defibrillator (ICD) with atrial lead to ensure continuous rhythm monitoring during follow up. At baseline, we will gather clinical and device data of patients. For AF prediction based on surface Electrocardiography (ECG), 24-h Holter ECG monitoring will be performed. After 6 months, we will assess the occurrence of AF during the study period via interrogation of PM/ICD. The resulting data will be used to develop algorithms including clinical, device and ECG data for prediction of the development of AF in individual patients. If possible, we will develop a risk score of high accuracy by combination of demographical, clinical and technical parameters of device patients. The resulting risk score could potentially help to facilitate the decision if anticoagulation is necessary in patients with either risk of AF or embolic stroke of unknown origin. Furthermore, Hayn et al. (AIT Austrian Institute of Technology) are currently developing algorithms to predict the occurrence of AF surface ECG data. It is an additional aim of this project to support the development of this algorithm in pacemaker and ICD patients and to increase the accuracy of AF prediction with clinical parameters and other parameters available to patients with implanted pacemaker (PM) or implanted cardioverter-defibrillator (ICD).

ELIGIBILITY:
Inclusion Criteria:

* Implanted pacemaker or implanted cardioverter defibrillator (ICD) with atrial lead
* CHADS-VASc Score of 2 or more
* Sinus rhythm or atrial paced rhythm
* Atrial stimulation rate 50% or less
* ModeSwitch rate 50% or less since last pacemaker interrogation

Exclusion Criteria:

* pacemaker or ICD malfunction
* atrial fibrillation (AF) at time of pacemaker / ICD interrogation
* AF during 24-hour Holter ECG monitoring
* permanent AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an implanted dual-chamber Pacemaker or an implantable cardioverter Defibrillator
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of atrial high rate episodes | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No